CLINICAL TRIAL: NCT06618755
Title: IMMANENCE - Intérêt d'un Suivi Sous Forme d'Entretiens Motivationnels spécifiques Post Hospitalisation Sur le Maintien de l'AbstiNENCE Durant l'année Suivant le Sevrage en Alcool
Brief Title: Motivational Interviews Post Hospitalisation on Maintaining AbstiNence for 1 Year après le Sevrage en Alcool
Acronym: IMMANENCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RECHMPL22_0564
Record Dates: First submitted 2024-09-24; First posted 2024-10-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Alcohol Use Disorder; Addiction; Alcohol Withdrawal; Motivational Interviews; Relapse
MeSH Terms: conditions — Alcoholism; Behavior, Addictive; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group : PSH (usual care) with motivational interviewing (Experimental): People randomised to the experimental group will have scheduled appointments to collect study data (monthly assessment). They will take part in an initial motivational interview to lay the foundations for the work that will be carried out throughout the follow-up period. Then, for 4 and a half months, a motivational interview will be scheduled every 14 days.
  Interventions: Other: Experimental group : PSH (usual care) with motivational interviewing
- Control group : PSH (usual care) (No Intervention): People randomised to the control group will have scheduled appointments for study-related data collection (monthly assessment), in addition to their routine care.

INTERVENTIONS:
Other: Experimental group : PSH (usual care) with motivational interviewing — The experimental group will begin follow-up after the 1st inclusion visit, during hospitalisation for withdrawal. The first motivational interview will take place 1 to 4 days before discharge from full hospitalisation. The following 10 motivational interviews will be held 2 weeks apart and will follow a framework based on the following objectives: to create a relationship of trust and an effective and lasting therapeutic alliance from the first interview; to create personalised objectives for the user, in line with their addictive pathology; to support the user as they modify, 'fail' and 'succeed' in achieving these objectives; to encourage the emergence and maintenance of the user's desire to change.
  Arms: Experimental group : PSH (usual care) with motivational interviewing

SUMMARY:
The aim of this clinical study is to evaluate the efficacy of reinforced inpatient aftercare versus usual care on the percentage of days of abstinence during the first year following withdrawal in adults with alcohol use disorders undergoing inpatient withdrawal. The hypothesis is that reinforced post-withdrawal follow-up, of the motivational interview type, during the first 4 months following hospitalisation, in addition to the usual care, would allow :

* Increase the percentage of days of abstinence in the year following withdrawal.
* Reduce the rate of relapse in the year following withdrawal.
* An increase in the cumulative and maximum duration of abstinence, an increase in motivation to maintain the change initiated and a reduction in the use of other substances in the year following withdrawal.
* A reduction in the impact of risk factors involved in the relapse process in the year following withdrawal.

All participants will have assessments to monitor their abstinence and consumption. In addition to their assessments, the experimental group will have motivational talks once every 15 days.

DETAILED DESCRIPTION:
In Europe, and particularly in France, there is a high level of alcohol consumption per capita (2.51 standard drinks/day/inhabitant in France in 2019). This consumption is not without risk, since 7% of all deaths in France in 2015 were attributable to alcohol, not to mention disabling pathologies and injuries. The treatment of alcohol addiction has many facets (social, neurological, psychological, behavioural, etc.) and involves a number of stages. One aspect that is particularly decisive in the consolidation phase of withdrawal (the phase following withdrawal when the risk of relapse is high) is the motivational dimension, which is widely described in the literature. Motivational Interviewing (MI) is a particularly effective tool for initiating and maintaining change. This tool, provided on a regular basis after discharge from hospital, helps to reinforce and maintain abstinence, a change initiated by users at the time of withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* With alcohol use disorders defined by at least 2 DSM-V criteria for at least 12 months).
* Being treated for withdrawal in hospital.
* With a goal of complete abstinence.
* With a means of communication (telephone).

Exclusion Criteria:

* Lack of understanding (written and spoken) of the French language.
* Breach of HC withdrawal contract, following failure to comply with the rules of the addictology service and somatic complications of addiction.
* Eviction from the department, discharge against medical advice during hospitalisation for withdrawal.
* Proven cognitive problems compromising understanding of the implications of the study and the proposed follow-up. proposed follow-up.
* Serious decompensated somatic pathology.
* Non-membership or non-beneficiaries of a national health insurance scheme.
* Person protected by law, under guardianship or curatorship.
* Not having signed free and informed consent to participate in the research.
* Simultaneous participation in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2028-01-13 (Estimated); Study Completion 2028-01-13 (Estimated)

PRIMARY OUTCOMES:
Percentage of days of abstinence over the 12 months following hospitalization for alcohol | From inclusion,once a month for 1 year
  The measures used for our main criterion will be declarative and collected on paper and by telephone every month in terms of the number of drinks per day. To facilitate data collection, the Timeline Follow Back method [30], developed by Sobell and also validated by telephone, will be used. This tool enables estimates of daily consumption of standard glasses to be collected retrospectively (for up to 12 months). The advantage of this method is that it reduces recall bias, since the participant can fill in a calendar from day to day and the data are collected every month.

SECONDARY OUTCOMES:
Relapse rates at 5 and 12 months | From inclusion,once a month for 1 year
  Percentage of patients who have relapsed (above WHO recommendations for low-risk drinking) at least once in the 5 and 12 months following hospitalisation for alcohol withdrawal. This relapse rate will be calculated on the basis of the consumption schedule collected using the method presented for the primary endpoint.
  As a reminder, the recommendations for lower-risk drinking are as follows:
  * No more than 10 standard drinks per week
  * No more than 2 standard drinks per day
  * Have days of the week when no alcohol is consumed.
Cumulative duration (in days) and maximum duration of abstinence over 5 and 12 months | Assessed 5 months after inclusion and 12 months after inclusion
  These cumulative and maximum periods of abstinence will be based on the consumption calendar collected using the Timeline Follow Back method.
Motivation to maintain abstinence | Assessed 0 month, 5 months and 12 months after inclusion
  Assessed using the Stages of Change Readiness and Treatment Eagerness Scale questionnaire
Craving felt | Assessed 0 month, 5 months and 12 months after inclusion
  Assessed using the Obsessive Compulsive Drinking Scale
Effectiveness of coping strategies | Assessed 0 month, 5 months and 12 months after inclusion
  Assessed using the Way og Coping Checklist questionnaire
Level of anxiety/depression | Assessed 0 month, 5 months and 12 months after inclusion
  Assessed using the Hospital Anxiety and Depression scale questionnaire
Sense of personal effectiveness | Assessed 0 month, 5 months and 12 months after inclusion
  Assessed using the Sherer General Self-Efficacy Scale
Use of other substances | Assessed 0 month, 5 months and 12 months after inclusion
  Collection of data declarative data on consumption and quantification in the previous month

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas RISDORFER DE ISSDENTZI, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided